CLINICAL TRIAL: NCT06271187
Title: Development of Innovative Modular 3D-Printed Dynamic Orthoses: Application Programs for Hand Function Facilitation in Patients With Stroke
Brief Title: Dynamic-orthosis Programs for Stroke Hand Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Jer-Hao Chang, Associate Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-110-507
Record Dates: First submitted 2024-01-27; First posted 2024-02-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic-orthosis training group (Experimental): Participants will undergo traditional occupational therapy (2-3 times per week, one hour per session, for a total of six weeks), supplemented with an additional home-based dynamic orthotic therapy program (five days per week, one hour per session, for six weeks). The style of the dynamic orthosis will be selected by the researchers based on the participants' movement performance and rehabilitation goals, and it will be adjusted or replaced as their abilities progress.
  Interventions: Device: Dynamic-orthosis; Other: Traditional stroke occupational therapy training
- Regular training group (Other): Participants will receive traditional occupational therapy (2-3 sessions per week, one hour per session, for a total of six weeks). The training program includes muscle strength training, reaching and grasping exercises, manual tone control, motor facilitation, and activities of daily living training. During the study period, participants will not wear any hand dynamic orthosis during training.
  Interventions: Other: Traditional stroke occupational therapy training

INTERVENTIONS:
Device: Dynamic-orthosis — Engaging in motion training at home with the use of dynamic orthoses.
  Arms: Dynamic-orthosis training group
Other: Traditional stroke occupational therapy training — Traditional post-stroke movement training arranged by an occupational therapist in a medical setting.

SUMMARY:
This study aims to investigate the training benefits of modular 3D printed dynamic orthoses on upper limb function in stroke survivors.

DETAILED DESCRIPTION:
This study is a randomized controlled intervention trial. Participants are recruited from two medical centers in Taiwan and undergo a continuous 6-week intervention for post-stroke movement rehabilitation. The control group receives traditional stroke occupational therapy rehabilitation. The experimental group, in addition to traditional treatment, supplements their therapy with the use of modular 3D printed dynamic orthoses developed by the research team for home training. Both groups undergo two effectiveness follow-up assessments, one month and two months after the intervention.

ELIGIBILITY:
Inclusion criteria:

1. Onset of stroke at least three months ago;
2. Upper limb Brunnstrom stage II~IV;
3. Shoulder can actively flex at least 45 degrees.

Exclusion criteria:

1. Affected hand has regained autonomous grasping function, able to grasp and release a tennis ball 10 times within 2 minutes;
2. Joint deformity or stiffness in the affected hand that prevents the use of the dynamic orthosis;
3. Diagnosis of other neurological disorders affecting motor control, such as neglect, Parkinson's disease, etc.;
4. Inability to follow therapist guidance;
5. Currently undergoing other specific treatments affecting motor function recovery (such as rTMS and BTX).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment- Upper Extremity | Pre-test(Week 0), post-test(Week 6), follow-up assessment（Week 10 & Week 14）
  The Fugl-Meyer Assessment-Upper Extremity (FMA-UE) is a specialized test designed for evaluating motor function in individuals post-stroke. It employs an ordinal scale to score 33 items related to upper limb movements, with a total score of 66 points. Each item reflects movements indicative of motor function in post-stroke hemiparetic patients, covering a range from proximal to distal joints.
  The FMA-UE has undergone extensive testing and has been found to possess excellent psychometric properties. It is considered an effective assessment tool for upper limb motor function, particularly suitable for chronic stroke patients with moderate to severe impairments.
Box and Block Test | Pre-test(Week 0), post-test(Week 6), follow-up assessment（Week 10 & Week 14）
  The Box and Block Test (BBT) is a tool used to assess manual dexterity, known for its short assessment time, simplicity, and ease of understanding. It exhibits excellent test-retest reliability (0.96) and inter-rater reliability (0.99). The test involves counting the number of cubes a person can move within one minute, with a higher quantity indicating better functionality. The size of the cubes is 2.5cm³, and there are a total of 150 cubes. Past research suggests a Minimal Clinically Important Difference (MCID) value of 5.5 cubes for the BBT.
Motor Activity Log | Pre-test(Week 0), post-test(Week 6), follow-up assessment（Week 10 & Week 14）
  The Motor Activity Log (MAL) is a questionnaire-based assessment that evaluates the amount of use (AOU) and quality of movement (QOM) of the affected side in daily activities. The scoring for amount of use ranges from 0 (never using the affected hand in the activity) to 5 (always using the affected hand in the activity). Quality of movement is scored from 0 (unable to use the affected hand) to 5 (movement quality comparable to pre-stroke). There are a total of 28 items in the assessment, recording the average scores for both amount of use and movement quality for each item. Previous research has demonstrated good construct validity for this scale, with a Minimal Clinically Important Difference (MCID) ranging from 1.0 to 1.1 points.

SECONDARY OUTCOMES:
Modified Ashworth scale | Pre-test(Week 0), post-test(Week 6), follow-up assessment（Week 10 & Week 14）
  The MAS (Modified Ashworth Scale) utilizes quick stretching to assess muscle tone, with testing conducted on the upper limb, specifically the hand, elbow, wrist, and fingers. For ease of statistical analysis, the scale is converted into numerical values ranging from 0 to 5, with lower scores indicating lower muscle tone.
Upper limb joint range of motion | Pre-test(Week 0), post-test(Week 6), follow-up assessment（Week 10 & Week 14）
  This study will use a goniometer to measure the upper limb joint range of motion in patients, including the shoulder, elbow, wrist, and fingers. The measurements encompass passive range of motion (PROM), active range of motion without wearing orthosis (AROM), and active-assisted range of motion with orthosis assistance (AAROM).

CONTACTS AND LOCATIONS:
Overall Officials: JERHAO CHANG, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No